CLINICAL TRIAL: NCT04010448
Title: A Phase 3 Double-blind, Randomized, Active Comparator-controlled, Group-sequential, Multinational Trial to Assess the Safety, Immunogenicity and Efficacy of a Trivalent Rotavirus P2-VP8 Subunit Vaccine in Prevention of Severe Rotavirus Gastroenteritis in Healthy Infants
Brief Title: A Trial to Assess the Safety, Immunogenicity and Efficacy of a Trivalent Rotavirus P2-VP8 Subunit Vaccine in Prevention of Severe Rotavirus Gastroenteritis in Healthy Infants in Africa and India
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PATH (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); SK Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CVIA 061
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Rotavirus Infection of Children
MeSH Terms: interventions — RIX4414 vaccine

STUDY DESIGN:
Intervention Model Description: Participating infants will be randomized 1:1 to receive either: 1) 90 µg of the TV P2-VP8 vaccine IM plus oral placebo, or 2) Rotarix® PO plus IM placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To maintain the blind, infants allocated to the TV P2-VP8 vaccine arm will receive both TV P2-VP8 IM as well as oral placebo vaccine, and infants allocated to receive Rotarix® will receive both Rotarix® PO and placebo IM.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TV P2-VP8 (Experimental)
  Interventions: Biological: TV P2-VP8
- Rotarix® (Active Comparator)
  Interventions: Biological: Rotarix

INTERVENTIONS:
Biological: TV P2-VP8 — 90 µg of the TV P2-VP8 vaccine IM plus oral placebo administered on study days 1, 29 and 57
  Arms: TV P2-VP8
Biological: Rotarix — Rotarix® PO plus IM placebo administered on study days 1, 29 and 57
  Arms: Rotarix®

SUMMARY:
The trial will be a multinational, randomized, double-blind, double-dummy, endpoint driven, group-sequential, active comparator-controlled study, in which participating infants will be randomized 1:1 to receive either: 1) 90 µg of the TV P2-VP8 vaccine IM plus oral placebo, or 2) Rotarix® per os (PO) plus IM placebo. Participants will receive three doses of TV P2-VP8/placebo IM and two doses of Rotarix®/placebo PO at monthly intervals starting at ≥6 to <8 weeks of age, administered concomitantly with EPI/UIP vaccines. To maintain the blind, infants allocated to the TV P2-VP8 vaccine arm will receive both TV P2-VP8 IM as well as oral placebo vaccine, and infants allocated to receive Rotarix® will receive both Rotarix® PO and placebo IM. Active surveillance for episodes of gastroenteritis (GE) will be conducted throughout the study, through weekly contact with participants' parents. Unsolicited AEs grade ≥ 2 through 28 days after the last study vaccination will be recorded in the study database, as will data for SAEs (including intussusception) throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants as established by medical history and clinical examination before entering the study
* Age: ≥6 and <8 weeks at the time of first study vaccination (42 days through 55 days old, inclusive, with the day after birth considered 1-day old)
* Parental/legal guardian's ability and willingness to provide written informed consent
* Intention of the participants' parents to remain in the area with the child during the study period

Exclusion Criteria:

* Acute disease at the time of first study vaccination - temporary exclusion
* Presence of fever on the day of first study vaccination (axillary temperature >37.6oC) - temporary exclusion
* Concurrent participation in another clinical trial throughout the entire timeframe for this study (participation in non-interventional observational study is allowed if there is no blood draw)
* Presence of severe malnutrition (weight-for-height z-score ≤-3SD median, per WHO published child growth standards) or any systemic disorder (cardiovascular, pulmonary, hepatic, renal, gastrointestinal, hematological, endocrine, immunological, dermatological, neurological, cancer or autoimmune disease) as determined by medical history and/or physical examination that would compromise the participant's health or is likely to result in nonconformance to the protocol
* History of premature birth (<37 weeks gestation) and/or birth weight of <2.5 kg
* History of congenital abdominal disorders, intussusception, or abdominal surgery
* Prior receipt of rotavirus vaccine
* Known sensitivity or allergy to any components of the study vaccine
* Contraindication to any EPI/UIP vaccine
* History of anaphylactic reaction
* Major congenital or genetic defect
* Parents not able, available or willing to accept active weekly follow-up by the study staff
* Receipt of any immunoglobulin therapy and/or blood products
* Nursing infants whose mother are receiving immunosuppressive biologicals
* History of chronic administration (defined as more than 14 days) of immunosuppressant medications, including corticosteroids (those on inhaled or topical steroids may be permitted to participate in the study)
* Any medical condition in the participant or parents that, in the judgment of the investigator, would interfere with or serves as a contraindication to protocol adherence or a parents' ability to give informed consent

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8200 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of laboratory confirmed cases of severe rotavirus gastroenteritis (SRVGE; any strain) | For cases with onset at least 2 weeks after 3rd study vaccination and onset at any time after first vaccination; for all events within the first 2 years of life
  SRVGE is defined by a Vesikari score of >11 (primary analysis to be performed once >99 cases are identified with onset at least 2 weeks after receipt of third study vaccination)
Number of serious adverse events (SAEs), including intussusception | Through 28 days after the last dose of study vaccine
Number of Adverse Events (AEs) > or = to grade 2 | Through 28 days after the last dose of study vaccine

SECONDARY OUTCOMES:
Number of laboratory confirmed cases of very severe rotavirus gastroenteritis (VSRVGE; any strain) | For cases with onset at least 2 weeks after 3rd study vaccination and onset at any time after first vaccination; for all events within the first 2 years of life
  VSRVGE is defined by a Vesikari score of >15
Number of P-type specific (P[4], P[6] and P[8]) laboratory confirmed cases of SRVGE and VSRGE | For cases with onset at least 2 weeks after 3rd study vaccination and onset at any time after first vaccination; for all events within the first 2 years of life
Number of laboratory confirmed cases of rotavirus gastroenteritis (any strain) of any severity | For cases with onset at least 2 weeks after 3rd study vaccination and onset at any time after first vaccination; for all events within the first 2 years of life
Number of laboratory confirmed cases hospitalized for RVGE (any severity) | For cases with onset at least 2 weeks after 3rd study vaccination and onset at any time after first vaccination; for all events within the first 2 years of life
Incidence of SRVGE and VSRVGE per 100 children-years | For cases with onset at least 2 weeks after 3rd study vaccination and onset at any time after first vaccination; for all events within the first 2 years of life

CONTACTS AND LOCATIONS:
Overall Officials: George Armah, PhD, Principal Investigator — Noguchi Memorial Institute for Medical Research, University of Ghana, Legon; Desiree Witte, MD, Principal Investigator — Malawi-Liverpool-Wellcome Trust (MLW) Clinical Research Programme; Roma Chilengi, MD, Principal Investigator — Centre for Infectious Disease Research in Zambia (CIDRZ), Lusaka
Locations (1):
- Centre for Infectious Disease Research in Zambia (CIDRZ), Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Summary results for primary and secondary objectives
Supporting Information: Study Protocol, SAP
Time Frame: Within 12 months of completion of study
Access Criteria: Researchers who provide a methodologically sound proposal may be provided access after Sponsor permission.

REFERENCES:
- [Derived] Tewari T, Armah G, Cunliffe NA, Chisenga CC, Witte D, Kukula V, Jere KC, Simuyandi M, Damanka S, Mwinjiwa E, Kazimbaya K, Atuguba F, Williams J, Chilengi R, Csedrik J, Gast C, Fix A, Cryz S. Safety, immunogenicity, and relative efficacy of a parenteral trivalent rotavirus subunit vaccine candidate (TV P2-VP8) in healthy Ghanaian, Malawian, and Zambian infants. Vaccine. 2026 Jan 5;70:128019. doi: 10.1016/j.vaccine.2025.128019. Epub 2025 Nov 29. PMID 41319434